CLINICAL TRIAL: NCT02976909
Title: Paclitaxel In Combination With Cisplatin and 5-fluorouracil(TPF) Induction Chemotherapy for Locally Advanced Borderline-resectable Esophageal Squamous Cell Carcinoma: A Phase II Clinical Trial
Brief Title: Efficacy and Safety of TPF Induction Chemotherapy for Borderline-resectable Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPF-1
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel+Cisplatin+5fluorouracil (Experimental): Patients will receive the following chemotherapy: Paclitaxel 135mg/m2 IV over 3 hours on Day 1; Cisplatin 75mg/m2 IV over 1 hours on Day 1; 5-FU 4g/m2 for 5 days continuous infusion from Day 1 to Day 5.
  Interventions: Drug: Paclitaxel+Cisplatin+5fluorouracil

INTERVENTIONS:
Drug: Paclitaxel+Cisplatin+5fluorouracil — Patients will receive the following chemotherapy: Paclitaxel 135mg/m2 IV over 3 hours on Day 1; Cisplatin 75mg/m2 IV over 1 hours on Day 1; 5-FU 4g/m2 for 5 days continuous infusion from Day 1 to Day 5.
  Other Names: Paclitaxel; Cisplatin; 5fluorouracil

SUMMARY:
This trial studies the efficacy and safty of paclitaxel in combination with cisplatin and 5-fluorouracil(TPF) induction chemotherapy for locally advanced borderline-resectable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common malignant tumors in China. In Asian countries, esophageal squamous carcinoma is the main pathological type of esophageal carcinoma. Prognosis of esophageal squamous carcinoma is usually poor and surgery is the only radical treatment. However, the optimal therapy pattern for local advanced esophageal carcinoma is still unclear. Part of the patients that clinical staging as T4 and with bulky lymph node metastasis are initially diagnosed as borderline-resectable, which means patients may be able to undergo R0 resection. However, for patients who are diagnosed as borderline-resectable esophageal carcinoma, there are still no sufficient studies implicate that how to improve R0 resection rate by convertion chemotherapy. Cisplatin in combination with 5-FU and docetaxel regimen(DCF) was reported as effective neoadjuvant chemotherapy in treating esophageal squamous carcinoma. However, studies also showed that the DCF regimen caused severe adverse reaction. The mechanism of paclitaxel is similar to docetaxel while with less adverse events than docetaxel. Based on the research situation mentioned above, the investigators decided to conduct a phase II clinical trial to further explore the efficacy and safety of paclitaxel in combination with cisplatin and 5-FU (TPF) induction chemotherapy for locally advanced borderline-resectable esophageal squamous carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be voluntary to the trial and provide with signed informed consent.
2. Male or female patients, age:18-70 years old
3. Confirmed by histology of thoracic esophageal squamous cell carcinoma without metastasis and diagnosed as boundary resectable by Multidisciplinary consultation, including cT4 and/or bulky lymphadenopathy that may invade nearby organs(such as the great vessels, trachea and heart, etc.)
4. Measurable or unmeasurable lesions according the RECIST 1.1 criteria.
5. No previous chemotherapy or radiotherapy.
6. Life expectancy ≥ 3 months.
7. ECOG PS 0-1.
8. Blood routine within 7 days：Hb ≥9g/L，NE ≥1.5×109/L，PLT ≥100×109/L；
9. Hepatic and renal function：TB <1.5 UNL， Cr< 1.5× UNL， AST / ALT < 2.5× UNL， ALP < 5.0 × UNL。
10. No severe complications such as active digestive tract hemorrhage, perforation, jaundice, gastrointestinal obstruction, non-cancerous fever > 38 ℃
11. Fertile patients should take effective contraceptive measures.
12. Patients should have good compliance and cooperate with the evaluation of efficacy and adverse events and follow-ups according to the research plan.

Exclusion Criteria:

1. Cervical esophageal carcinoma.
2. Known severe hypersensitivity to drugs in the regimen.
3. Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment(with the exception of nonmelanoma skin cancer or cervical carcinoma in situ).
4. Evidence of serious heart disease, including recorded history of congestive heart-failure, uncontrolled serious arrhythmia, angina that needs treatment of drugs, clinical diagnosed cardiac valve disease, history of serious myocardial infarction and intractable hypertension.
5. Evidence of chronic diarrhea(≥4 times/day) or renal dysfunction.
6. Evidence of active infection or active epidemic disease.
7. Psychiatric illness that would prevent the patient from giving informed consent
8. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | following resection for up to 36 months
  The rate of R0 resection

SECONDARY OUTCOMES:
pathologic complete response rate | following resection for up to 36 months
  The rate of pathologic complete response following surgery
OS | for up to 36 months
  the duration from enrollment to the patient's death (all causes)
PFS | for up to 36 months
  the duration from enrollment to tumour progression or the patient's death (all causes) (whichever comes first)
Adverse envents | for up to 12 months
  Incidence of AEs and SAEs during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-hong Li, MD, Ph D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wu JD, Wang ZQ, Li QQ, Li ZC, Ren C, Wang DS, Chen JY, Tan Q, Li YH, Yang H. A 3-Year Survival Update from a Phase 2 Study of Paclitaxel Plus Cisplatin and 5-Fuorouracil Induction Chemotherapy for Locally Advanced Borderline-Resectable Esophageal Squamous Cell Carcinoma: The NEOCRTEC-1601 Clinical Trial. Ann Surg Oncol. 2024 Feb;31(2):838-846. doi: 10.1245/s10434-023-14513-0. Epub 2023 Nov 2. PMID 37919448
- [Derived] Wang Z, Hu M, Hu Y, Li Q, Wu J, Fong WP, Ren C, Wang D, Tan Q, Yang H, Li Y. Paclitaxel plus cisplatin and 5-fluorouracil induction chemotherapy for locally advanced borderline-resectable esophageal squamous cell carcinoma: a phase II clinical trial. Esophagus. 2022 Jan;19(1):120-128. doi: 10.1007/s10388-021-00864-8. Epub 2021 Jul 28. PMID 34319435